CLINICAL TRIAL: NCT00881946
Title: A Phase I, Open-Label, Two-Stage Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of the Oral AKT Inhibitor GSK2110183 in Subjects With Any Hematologic Malignancy
Brief Title: Repeat Dose Safety Study for Compound to Treat Hematologic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Accenture (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PKB112835
Record Dates: First submitted 2009-03-20; First posted 2009-04-15 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Hematologic Malignancies
Keywords: chronic lymphocytic leukemia; aggressive lymphoma; non-Hodgkin's lymphoma; Hodgkin's lymphoma; chronic myelogenous leukemia; multiple myeloma; acute lymphoblastic leukemia; acute myeloid leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2119183 (Experimental)
  Interventions: Drug: GSK21110183

INTERVENTIONS:
Drug: GSK21110183 — Starting Dose = 25mg once daily with dose escalation until unacceptable toxicity develops

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of repeat doses of compound GSK2110183 in subjects with hematologic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is provided.
2. Male or female who is at least 18 years of age or older.
3. Histologically- or cytologically-confirmed diagnosis of a hematologic malignancy - that has relapsed or is refractory after standard therapy, AND that is not associated with human immunodeficiency virus (HIV) infection or solid organ transplant, including:

   * chronic lymphocytic leukemia (CLL),
   * chronic myelogenous leukemia (CML),
   * multiple myeloma (MM),
   * non-Hodgkin's lymphoma (NHL),
   * Hodgkin's lymphoma, or
   * Other hematologic malignancy excluding:
   * acute leukemia of any type
   * CML blast crisis
   * myelodysplastic syndrome (MDS)
   * myelofibrosis
4. Performance Status score of 0 and 1 according to the Eastern Cooperative Oncology Group (ECOG) scale
5. Able to swallow and retain oral medication.
6. Fasting serum glucose < 126 mg/dL (<7 mmol/L).
7. Male subjects with a female partner of childbearing potential must have had a prior vasectomy or agree to use adequate contraception from the time of the first dose of study drug until three months after the last dose of study drug.
8. A female subject is eligible to participate if she is of:

   * Non-childbearing potential
   * Child-bearing potential, has a negative serum pregnancy test during the screening period, and agrees to use adequate contraception from screening until four weeks after the last dose of study drug.
9. Adequate organ system function

Exclusion Criteria:

1. Chemotherapy, radiotherapy, or immunotherapy within 28 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of study drug.
2. Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is longer, preceding the first dose of study drug.
3. Current use of a prohibited medication or requires any of these medications during treatment with study drug.
4. Current use of anticoagulants at therapeutic levels within seven days prior to the first dose of study drug, including warfarin, low molecular weight heparin and direct thrombin inhibitors. Low dose (prophylactic) anticoagulants are permitted provided that subject's PT and PTT meet entry criteria.
5. Current use of any anti-platelet agent (e.g. dipyridamole, clopidogrel) other than aspirin (81 mg daily).
6. Presence of active gastrointestinal disease or other condition that could affect gastrointestinal absorption (e.g. malabsorption syndrome) or predispose subject to gastrointestinal ulceration.
7. Any major surgery within the last four weeks.
8. Unresolved toxicity (except alopecia) Grade 2 from previous anti-cancer therapy unless agreed to by a Medical Monitor and the Investigator
9. Previously diagnosed diabetes mellitus (Type 1 or 2).
10. Current use of oral corticosteroids, with the exception of inhaled or topical corticosteroids.
11. Any serious or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject safety or with obtaining informed consent.
12. Symptomatic or untreated central nervous system (CNS) involvement by the hematologic malignancy (including primary CNS lymphoma).
13. Evidence of severe or uncontrolled systemic diseases
14. Known infection with HIV, HBV or HCV.
15. QTc interval ≥ 470 msecs.
16. Other clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular (AV) block.
17. History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within the past six months.
18. Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
19. Pregnant or lactating female.
20. Active drug or alcohol abuse.
21. History of sensitivity to heparin or heparin-induced thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Physical exam | Screening, Days -3, 8, At the start of each additional Cycle
Electrocardiogram (ECG) | Days -3, -2, -1, 8, 15, At the start of each additional Cycle
Vital signs | Screening, Days -3, -2, -1, 8, 15, At the start of each additional Cycle
Transthoracic Echocardiogram (TTE)/Multiple Gated Acquisition (MUGA) Scans | Screening, Additionally as needed
Clinical Laboratory assessments | Screening, Days -3, 1, 8, 15, At the start of each additional Cycle
ECOG Peformance Status | Screening, Days -3, 8, At the start of each additional Cycle
PK - Maximum observed plasma concentraion (Cmax) | Days -3, -2, -1, 8, 15
PK - time to Cmax [tmax] (Maximum observed plasma concentration) | Days -3, -2, -1, 8, 15
PK - Area under the plasma concentration-time curve (AUC(0-t)) | Days -3, -2, -1, 8, 15
PK - Apparent terminal phase elimination rate constant | Days -3, -2, -1, 8, 15
PK - Apparent terminal phase half-life (t1/2) | Days -3, -2, -1, 8, 15
PK - oral clearance (CL/F) | Days -3, -2, -1, 8, 15

SECONDARY OUTCOMES:
Metabolite Profiling | Days -3, 8

CONTACTS AND LOCATIONS:
Overall Officials: S. Jamie Freedman, MD, PhD, Study Director
Locations (4):
- Australia (2):
  - Prince of Wales Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Spencer A, Yoon SS, Harrison SJ, Morris SR, Smith DA, Brigandi RA, Gauvin J, Kumar R, Opalinska JB, Chen C. The novel AKT inhibitor afuresertib shows favorable safety, pharmacokinetics, and clinical activity in multiple myeloma. Blood. 2014 Oct 2;124(14):2190-5. doi: 10.1182/blood-2014-03-559963. Epub 2014 Jul 29. PMID 25075128